CLINICAL TRIAL: NCT00892437
Title: A Phase 2, Randomized, Double-Blinded Study of the Safety and Efficacy of GS-9350-boosted Atazanavir (ATV/GS-9350) Compared to Ritonavir-boosted Atazanavir (ATV/r) in Combination With Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Brief Title: Safety and Efficacy of Cobicistat-boosted Atazanavir Compared to Ritonavir-boosted Atazanavir in Combination With Emtricitabine/Tenofovir Disoproxil Fumarate in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-216-0105
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Results first posted 2014-10-28 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: HIV-1 Infection
Keywords: HIV; HIV-1; Antiretroviral Treatment-Naive
MeSH Terms: interventions — Cobicistat; Ritonavir; Atazanavir Sulfate; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATV+COBI+FTC/TDF (Experimental): COBI + RTV placebo +ATV+FTC/TDF for 48 weeks
  Interventions: Drug: COBI; Drug: ATV; Drug: FTC/TDF; Drug: RTV placebo
- ATV+RTV+FTC/TDF (Active Comparator): RTV + COBI placebo +ATV+FTC/TDF for 48 weeks
  Interventions: Drug: RTV; Drug: ATV; Drug: FTC/TDF; Drug: COBI placebo

INTERVENTIONS:
Drug: COBI — Cobicistat (COBI) 150 mg tablet administered orally once daily
  Other Names: Tybost®; GS-9350
  Arms: ATV+COBI+FTC/TDF
Drug: RTV — Ritonavir (RTV) 100 mg soft gelatin capsule administered orally once daily
  Other Names: Norvir®
  Arms: ATV+RTV+FTC/TDF
Drug: ATV — Atazanavir (ATV) 300 mg capsule administered orally once daily
  Other Names: Reyataz®
Drug: FTC/TDF — Emtricitabine (FTC) 200 mg/tenofovir disoproxil fumarate (TDF) 300 mg fixed-dose combination tablet administered orally once daily
  Other Names: Truvada®
Drug: COBI placebo — Placebo to match COBI administered orally once daily
  Arms: ATV+RTV+FTC/TDF
Drug: RTV placebo — Placebo to match RTV administered orally once daily
  Arms: ATV+COBI+FTC/TDF

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of a regimen containing cobicistat-boosted atazanavir (ATV+COBI) plus emtricitabine/tenofovir disoproxil fumarate (Truvada®; FTC/TDF) versus ritonavir-boosted atazanavir (ATV+RTV) plus FTC/TDF in HIV-1 infected, antiretroviral treatment-naive adults.

Participants will be randomized in a 2:1 ratio. Randomization will be stratified by HIV-1 RNA level (≤ 100,000 copies/mL or > 100,000 copies/mL) at screening. After Week 48, participants will continue to take their blinded study drug and attend visits every 12 weeks until treatment assignments are unblinded, at which point all participants will return for an unblinding visit and be given the option to participate in an open-label rollover extension and receive ATV+COBI+FTC/TDF until COBI tablets become commercially available, or until Gilead Sciences elects to terminate the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent form
* Plasma HIV-1 RNA levels ≥ 5,000 copies/mL
* No prior use of any approved or experimental anti-HIV drug
* Normal ECG (or if abnormal, determined by the investigator to be not clinically significant)
* Adequate renal function (estimated glomerular filtration rate ≥ 80 mL/min according to the Cockcroft-Gault formula)
* Hepatic transaminases ≤ 2.5 × upper limit of normal
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function (absolute neutrophil count ≥ 1000/mm^3; platelets ≥ 50,000/mm^3; hemoglobin ≥ 8.5 g/dL)
* Cluster of differentiation 4 (CD4) cell count > 50 cells/µL
* Serum amylase ≤ 1.5 × ULN (subjects with serum amylase >1.5 × ULN remained eligible if serum lipase is ≤ 1.5 × ULN)
* Normal thyroid-stimulating hormone
* Negative serum pregnancy test (females of childbearing potential only)
* Males and females of childbearing potential must agree to utilize highly effective contraception methods from screening throughout the duration of study treatment and for 30 days following the last dose of study drugs
* Age ≥ 18 years
* Life expectancy ≥ 1 year

Exclusion Criteria:

* New AIDS-defining condition diagnosed within the 30 days prior to screening
* Documented drug resistance to nucleoside or nucleotide reverse transcriptase inhibitors (NRTIs), nonnucleoside reverse transcriptase inhibitors (NNRTIs), or primary PI resistance mutation(s)
* Hepatitis B surface antigen positive
* Hepatitis C antibody positive
* Participants experiencing cirrhosis
* Participants experiencing ascites
* Participants experiencing encephalopathy
* Females who are breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Vaccinated within 90 days of study dosing
* History or family history of Long QT Syndrome or have a family history of sudden cardiac death or unexplained death in an otherwise healthy individual under the age of 30 years
* Presence or history of cardiovascular disease, cardiomyopathy, and/or cardiac conduction abnormalities
* Prolonged QTcF (QT interval corrected for heart rate using Fridericia's formula) interval at screening (eg, a prolongation of the QTcF interval of greater than 450 msec for males and greater than 470 msec for females)
* PR interval greater than or equal to 200 msec or less than or equal to 120 msec on ECG at screening
* QRS greater than or equal to 120 msec on ECG at screening
* Implanted defibrillator or pacemaker
* Subjects receiving ongoing therapy with any disallowed medications
* Current alcohol or substance use judged to potentially interfere with subject study compliance
* History of or ongoing malignancy (including untreated carcinoma in-situ) other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Participation in any other clinical trial without prior approval
* Medications contraindicated for use with ATV, RTV, FTC, or TDF
* Any known allergies to the excipients of ATV capsules, RTV capsules, COBI tablets or FTC/TDF tablets
* Any other clinical condition or prior therapy that would make the subject unsuitable for the study or unable to comply with the dosing requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Fordyce, MD, Study Chair — Gilead Sciences
Locations (31):
- United States (31):
  - Southwest Center for HIV/AIDS, Phoenix, Arizona
  - Health for Life Clinic, PLLC, Little Rock, Arkansas
  - AIDS Healthcare Foundation-Research Center, Beverly Hills, California
  - The Living Hope Foundation, Long Beach, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - David J. Shamblaw, MD Inc., San Diego, California
  - Metropolis Medical, San Francisco, California
  - Denver Infectious Disease Consultants, PLLC, Denver, Colorado
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Capital Medical Associates PC, Washington D.C., District of Columbia
  - Gary Richmond, MD, PA, Inc., Fort Lauderdale, Florida
  - Wohlfeiler, Piperato and Associates, LLC, Miami Beach, Florida
  - ValuehealthMD, LLC, Orlando, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta (IDSA), Decatur, Georgia
  - Northstar Medical Center, Chicago, Illinois
  - Chase Brexton Health Services, Inc., Baltimore, Maryland
  - Be Well Medical Center, Berkley, Michigan
  - Central West Healthcare, St Louis, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Saint Michael's Medical Center, Newark, New Jersey
  - Southwest C.A.R.E. Center, Santa Fe, New Mexico
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Nicholaos Bellos, MD, PA, Dallas, Texas
  - AIDS Arms/ Peabody Health Center, Dallas, Texas
  - Gordon E. Crofoot, MD, PA, Houston, Texas
  - Therapeutic Concepts, P.A., Houston, Texas
  - TribalMed, Seattle, Washington

REFERENCES:
- [Result] Elion R, Cohen C, Gathe J, Shalit P, Hawkins T, Liu HC, Mathias AA, Chuck SL, Kearney BP, Warren DR; GS-US-216-0105 Study Team. Phase 2 study of cobicistat versus ritonavir each with once-daily atazanavir and fixed-dose emtricitabine/tenofovir df in the initial treatment of HIV infection. AIDS. 2011 Sep 24;25(15):1881-6. doi: 10.1097/QAD.0b013e32834b4d48. PMID 21811136

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated in 32 study centers in the United States. The first participant was screened on 04 May 2009, and the last study visit occurred on 15 January 2015.
Pre-assignment Details: 137 participants were screened.
Groups:
- ATV+COBI+FTC/TDF: Randomized Phase: Cobicistat (COBI) 150 mg + ritonavir (RTV) placebo + atazanavir (ATV) 300 mg + emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) (200/300 mg) once daily
  Open-Label Extension Phase: COBI 150 mg + ATV 300 mg + FTC/TDF (200/300 mg) once daily
- ATV+RTV+FTC/TDF: Randomized Phase: RTV 100 mg + COBI placebo + ATV 300 mg + FTC/TDF (200/300 mg) once daily
  Open-Label Extension Phase: COBI 150 mg + ATV 300 mg + FTC/TDF (200/300 mg) once daily
Period: Randomized Phase
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Started | 56 | 29
Randomized and Treated | 50 | 29
Completed | 45 | 24
Not Completed | 11 | 5
Not completed — Randomized but not treated | 6 | 0
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 1 | 3
Not completed — Investigator's Discretion | 1 | 0
Not completed — Withdrew Consent | 1 | 0
Period: Open-Label Extension Phase
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Started | 44 (1 participant completed the randomized phase but did not enter the open-label extension phase.) | 19 (5 participants completed the randomized phase but did not enter the open-label extension phase.)
Completed | 32 | 15
Not Completed | 12 | 4
Not completed — Adverse Event | 4 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Investigator's Discretion | 1 | 0
Not completed — Withdrew Consent | 3 | 1

BASELINE CHARACTERISTICS:
Population: ITT Analysis Set: participants who were randomized and received at least one dose of study drug.
Groups:
- ATV+COBI+FTC/TDF: Randomized Phase: COBI 150 mg + RTV placebo + ATV 300 mg + FTC/TDF (200/300 mg) once daily
  Open-Label Extension Phase: COBI 150 mg + ATV 300 mg + FTC/TDF (200/300 mg) once daily
- Total: Total of all reporting groups
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF | Total
Number analyzed (Participants) | 50 | 29 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (9.6) | 34 (10.1) | 36 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 47 | 25 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 43 | 24 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 2 | 2
  Black | 18 | 9 | 27
  White | 31 | 16 | 47
  Other | 1 | 2 | 3
HIV-1 RNA [Mean (Standard Deviation); unit: log_10 copies/mL] | 4.56 (0.657) | 4.69 (0.530) | 4.61 (0.614)
HIV-1 RNA Category [Number; unit: participants]
  ≤ 100,000 copies/mL | 38 | 18 | 56
  > 100,000 copies/mL | 12 | 11 | 23
Cluster of differentiation (CD4) Cell Count [Mean (Standard Deviation); unit: cells/uL] | 365 (201.3) | 343 (178.1) | 357 (192.2)
CD4 Cell Count Category [Number; unit: participants]
  ≤ 50 cells/μL | 1 | 1 | 2
  51 to ≤ 200 cells/μL | 9 | 6 | 15
  201 to ≤ 350 cells/μL | 16 | 7 | 23
  351 to ≤ 500 cells/μL | 17 | 11 | 28
  > 500 cells/μL | 7 | 4 | 11
HIV Disease Status [Number; unit: participants]
  Asymptomatic | 41 | 25 | 66
  Symptomatic HIV Infections | 1 | 1 | 2
  AIDS | 8 | 3 | 11
Chronic Hepatitis B Infection Status [Number; unit: participants]
  Negative | 50 | 29 | 79
  Positive | 0 | 0 | 0
Chronic Hepatitis C Infection Status [Number; unit: participants]
  Negative | 50 | 29 | 79
  Positive | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the missing = failure method, where participants with missing data were considered to have failed to achieve the endpoint.
Time Frame: Week 24
Population: ITT Analysis Set: participants who were randomized and received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Number analyzed (Participants) | 50 | 29
percentage of participants | 84.0 | 89.7
Statistical Analysis 1: Comparison: ATV+COBI+FTC/TDF vs ATV+RTV+FTC/TDF; A total planned sample size of 75 subjects had 26% power to evaluate noninferiority with respect to the response rate of HIV-1 RNA < 50 copies/mL at Week 24 if a response rate of 84% for both arms and a noninferiority margin of 0.12 were assumed; Test type: Non-Inferiority or Equivalence — Null hypothesis: the response rate in the ATV+COBI+FTC/TDF group was at least 12% worse than in the ATV+RTV+FTC/TDF group; alternative hypothesis: the response rate in the ATV+COBI+FTC/TDF group was less than 12% worse than that in the ATV+RTV+FTC/TDF group. ATV+COBI+FTC/TDF was noninferior if the lower bound of the 2-sided 95% confidence interval (CI) of the baseline HIV-1 RNA stratum-weighted difference (COBI group - RTV group) in the response rate at Week 24 was greater than -12%; Difference in percentages = -7.4, 95% CI 2-sided [-24.6 to 9.9] — Difference in percentages of success and its 95% confidence interval (CI) were calculated based on baseline HIV-1 RNA stratum-adjusted Mantel-Haenszel (MH) proportion

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the missing = failure method.
Time Frame: Week 48
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Number analyzed (Participants) | 50 | 29
percentage of participants | 82.0 | 89.7
Statistical Analysis 1: Comparison: ATV+COBI+FTC/TDF vs ATV+RTV+FTC/TDF; Test type: Non-Inferiority or Equivalence — The null hypothesis was that the response rate in the ATV+COBI+FTC/TDF group was at least 12% worse than the response rate in ATV+RTV+FTC/TDF group; the alternative hypothesis was that the response rate in the ATV+COBI+FTC/TDF group was less than 12% worse than that in the ATV+RTV+FTC/TDF group; Difference in percentages = -8.3, 95% CI 2-sided [-25.9 to 9.4] — Difference in percentages of success and its 95% CI were calculated based on baseline HIV-1 RNA stratum-adjusted MH proportion

3. Secondary Outcome: Change From Baseline in HIV-1 RNA at Week 24
Description: The change from baseline in log_10 HIV-1 RNA at Week 24 was analyzed.
Time Frame: Baseline to Week 24
Population: Participants in the ITT Analysis Set with available change data at Week 24 were analyzed.
Measure: Mean (Standard Deviation); unit: log_10 copies/mL
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Number analyzed (Participants) | 46 | 27
log_10 copies/mL | -2.80 (0.619) | -2.97 (0.707)
Statistical Analysis 1: Comparison: ATV+COBI+FTC/TDF; Test type: Superiority or Other; p = 0.87, ANOVA — P-values were obtained from an ANOVA model including baseline HIV-1 RNA category in the model; Difference in least squares mean (LSM) = -0.02, 95% CI 2-sided [-0.25 to 0.22] — The difference in least squares mean (LSM) and its 95% CI were computed using ANOVA model, including baseline HIV-1 RNA category in the model

4. Secondary Outcome: Change From Baseline in HIV-1 RNA at Week 48
Description: The change from baseline in log_10 HIV-1 RNA at Week 48 was analyzed.
Time Frame: Baseline to Week 48
Population: Participants in the ITT Analysis Set with available change data at Week 48 were analyzed.
Measure: Mean (Standard Deviation); unit: log_10 copies/mL
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Number analyzed (Participants) | 46 | 27
log_10 copies/mL | -2.79 (0.678) | -2.96 (0.765)
Statistical Analysis 1: Comparison: ATV+COBI+FTC/TDF vs ATV+RTV+FTC/TDF; Test type: Superiority or Other; p = 0.82, ANOVA — P-values were obtained from an ANOVA model including baseline HIV-1 RNA category in the model; Difference in LSM = -0.03, 95% CI 2-sided [-0.30 to 0.23] — The difference in LSM and its 95% CI were computed using ANOVA model, including baseline HIV-1 RNA category in the model

5. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 24
Description: The change from baseline in CD4 cell count at Week 24 was analyzed.
Time Frame: Baseline to Week 24
Population: Participants in the ITT Analysis Set with available change data at Week 24 were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Number analyzed (Participants) | 46 | 26
cells/μL | 200 (164.6) | 202 (115.1)
Statistical Analysis 1: Comparison: ATV+COBI+FTC/TDF vs ATV+RTV+FTC/TDF; Test type: Superiority or Other; p = 0.78, ANOVA — P-values were obtained from an ANOVA model including baseline HIV-1 RNA category in the model; Difference in LSM = 10, 95% CI 2-sided [-63 to 84] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48
Description: The change from baseline in CD4 cell count at Week 48 was analyzed.
Time Frame: Baseline to Week 48
Population: Participants in the ITT Analysis Set with available change data at Week 48 were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF
Number analyzed (Participants) | 46 | 27
cells/μL | 243 (186.5) | 213 (168.2)
Statistical Analysis 1: Comparison: ATV+COBI+FTC/TDF vs ATV+RTV+FTC/TDF; Test type: Superiority or Other; p = 0.29, ANOVA — P-values were obtained from an ANOVA model including baseline HIV-1 RNA category in the model; Difference in LSM = 47, 95% CI 2-sided [-41 to 134] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline through end of study (average of 169.9 weeks; maximum of 286 weeks)
Groups:
- ATV+COBI+FTC/TDF: For the reporting of Adverse Events, this group includes participants who were randomized to receive COBI 150 mg + RTV placebo + ATV 300 mg + FTC/TDF (200/300 mg) once daily in the randomized phase, and were analyzed from Baseline to Week 60.
- ATV+RTV+FTC/TDF: For the reporting of Adverse Events, this group includes participants who were randomized to receive RTV 100 mg+COBI placebo+ATV 300 mg+FTC 200 mg/TDF 300 mg once daily in the randomized period, and were analyzed from Baseline to Week 60.
- All ATV+COBI+FTC/TDF: The All ATV+COBI+FTC/TDF Safety Analysis Set included all participants who received at least 1 dose of COBI 150 mg + ATV 300 mg + FTC/TDF (200/300 mg) in the randomized phase or in the open-label extension phase. Adverse event data presented in this group include the following: Adverse events collected from participants who were initially randomized to the double-blind ATV+COBI+FTC/TDF group while they received double-blind ATV+COBI+FTC/TDF during the randomized phase and open-label ATV+COBI+FTC/TDF during the extension phase; adverse events collected from the open-label ATV+COBI+FTC/TDF extension phase only from the participants who were initially randomized to the ATV+RTV+FTC/TDF group during the randomized phase. Adverse event data collected up to Week 286 are presented in this entry.
Arm/Group | ATV+COBI+FTC/TDF | ATV+RTV+FTC/TDF | All ATV+COBI+FTC/TDF
Serious Adverse Events (participants affected / at risk) | 2/50 | 2/29 | 13/69
Other Adverse Events (participants affected / at risk) | 34/50 | 23/29 | 54/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATV+COBI+FTC/TDF (N=50) | ATV+RTV+FTC/TDF (N=29) | All ATV+COBI+FTC/TDF (N=69)
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Accidental death (General disorders) | 0 | 0 | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 2
Meningitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Prostate cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATV+COBI+FTC/TDF (N=50) | ATV+RTV+FTC/TDF (N=29) | All ATV+COBI+FTC/TDF (N=69)
Ocular icterus (Eye disorders) | 7 | 4 | 9
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 5 | 9 | 11
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 2 | 10
Chest pain (General disorders) | 3 | 0 | 5
Fatigue (General disorders) | 4 | 5 | 8
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 0 | 5
Jaundice (Hepatobiliary disorders) | 2 | 2 | 2
Acute sinusitis (Infections and infestations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 4 | 4 | 13
Cellulitis (Infections and infestations) | 1 | 0 | 4
Folliculitis (Infections and infestations) | 1 | 4 | 2
Gonorrhoea (Infections and infestations) | 1 | 1 | 5
Influenza (Infections and infestations) | 0 | 2 | 5
Nasopharyngitis (Infections and infestations) | 0 | 3 | 5
Pharyngitis (Infections and infestations) | 2 | 1 | 4
Sinusitis (Infections and infestations) | 5 | 3 | 11
Syphilis (Infections and infestations) | 2 | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 6 | 2 | 11
Weight increased (Investigations) | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 6
Dizziness (Nervous system disorders) | 2 | 3 | 5
Headache (Nervous system disorders) | 3 | 0 | 8
Sinus headache (Nervous system disorders) | 3 | 0 | 3
Anxiety (Psychiatric disorders) | 3 | 3 | 8
Depression (Psychiatric disorders) | 5 | 4 | 9
Insomnia (Psychiatric disorders) | 5 | 2 | 11
Nephrolithiasis (Renal and urinary disorders) | 3 | 0 | 5
Erectile dysfunction (Reproductive system and breast disorders) | 4 | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 10
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 5

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years